CLINICAL TRIAL: NCT00518726
Title: A Phase II, Open Label, Uncontrolled, Multi Center Study to Evaluate Safety and Immunogenicity of an Adjuvanted Influenza Vaccine Surface Antigen, Inactivated, Formulation 2007-2008, When Administered to Non-Elderly Adult and Elderly Subjects
Brief Title: Safety and Immunogenicity of a Commercially Available Influenza Vaccine (Formulation 2007/2008) When Administered to NON Elderly AND Elderly Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V71P5S; 2007-000963-28
Record Dates: First submitted 2007-08-20; First posted 2007-08-21 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Influenza
Keywords: Adjuvanted Influenza Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Antigens, Surface; Influenza Vaccines

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Biological: Surface Antigen, Inactivated, Adjuvanted, Influenza Vaccine, Formulation 2007-2008

INTERVENTIONS:
Biological: Surface Antigen, Inactivated, Adjuvanted, Influenza Vaccine, Formulation 2007-2008 — seasonal influenza vaccine 15ug

SUMMARY:
To evaluate the antibody response to each influenza vaccine antigen when administering a single dose to subjects aged > 18 years

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age or older

Exclusion Criteria:

* any serious disease such as cancer, autoimmune disease, advanced arteriosclerotic disease or complicated diabetes mellitus, chronic obstructive pulmonary disease (COPD) that requires oxygen therapy, acute or progressive hepatic disease, acute or progressive renal disease, congestive heart failure and bleeding diathesis or conditions associated with prolonged bleeding time hypersensitivity to eggs, chicken protein, chicken feathers, influenza viral protein, neomycin or polymyxin or any other component of the vaccine history of neurological symptoms or signs, or anaphylactic shock following administration of any vaccine known or suspected (or high risk of developing) impairment/alteration of immune function within the past 7 days, any acute disease or infections requiring systemic antibiotic or antiviral therapy fever within the past 3 days.No women in breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2007-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Safety and immunogenicity of seasonal inactivated, influenza vaccine, formulation 2007-2008, when administered to non-elderly adult and elderly subjects

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (3):
- Italy (3):
  - Dipartimento di Medicina e Scienze dell'Invecchiamento, Università G. D'Annunzio, Via Dei Vestini, Chieti
  - Ufficio Igiene e Sanità Pubblica di Lanciano, ASL Lanciano - Vasto sede legale, Via S. Spaventa, 37, Lanciano, Chieti
  - Presidio Distrettuale No. 8 Azienda Sanitaria USL 7 di Siena, Siena